CLINICAL TRIAL: NCT00956878
Title: Storage and Analysis of Patient Blood-samples for Cancer Pain Research
Brief Title: Cancer Pain Single Nucleotide Polymorphisms (SNPs)
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Joost LM Jongen, Dr. J.L.M. Jongen, MD, PhD, Erasmus Medical Center
Other Study IDs: MEC2008-166
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Cancer; Pain
Keywords: Cancer; Pain; SNP
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer Pain Patients

SUMMARY:
Cancer pain is common in advanced cancer patients. Opioids are the mainstay of treatment in cancer pain. Responsiveness to and tolerability of opioids is, amongst others, determined by small variations in human DNA. Using blood samples from clinically well-defined cancer pain patients, the investigators are going to analyze single nucleotide polymorphisms (SNPs) in genes that are known to be involved in responsiveness to opioids and sensitivity to pain.

ELIGIBILITY:
Inclusion Criteria:

* Cancer pain patients

Exclusion Criteria:

* Patients not able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer pain patients in a large university hospital
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2008-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
correlation between pain SNPs and equianalgesic opioid requirement | timepoint at blood sample
  candidate SNP analysis

CONTACTS AND LOCATIONS:
Overall Officials: Joost L Jongen, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Centrumlocatie en Daniel den Hoed, Rotterdam, South Holland, Netherlands

REFERENCES:
- See also: Related Info — http://www.erasmusmc.nl/neurologie